CLINICAL TRIAL: NCT03780309
Title: Using the Immediate Blood Pressure Benefits of Exercise to Improve Exercise Adherence Among Adults With Hypertension
Brief Title: Postexercise Hypotension and Exercise Adherence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Connecticut (Other)
Collaborators: Hartford Hospital (Other)
Responsible Party: Principal Investigator, Linda Pescatello, Board of Trustees Distinguished Professor, University of Connecticut
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H15-277HHC
Record Dates: First submitted 2018-12-11; First posted 2018-12-19 (Actual); Last update posted 2024-05-13 (Actual); Status verified 2024-05

CONDITIONS: Hypertension
Keywords: antihypertensive lifestyle therapy; positive outcome expectations; postexercise hypotension; self-efficacy; self-management
MeSH Terms: conditions — Hypertension; Post-Exercise Hypotension

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EXERCISE (Active Comparator): Participants participated in a the exercise training program and engaged in exercise self-monitoring.
  Interventions: Behavioral: Exercise Self-Monitoring
- EXERCISE+PEH (Experimental): Participants participated in the exercise training program and engaged in exercise self-monitoring and blood pressure self-monitoring (daily and before and after exercise).
  Interventions: Behavioral: Exercise Self-Monitoring; Behavioral: Blood Pressure Self-Monitoring

INTERVENTIONS:
Behavioral: Exercise Self-Monitoring — Participants engaged in exercise self-monitoring utilizing a traditional calendar recording method and heart rate monitor.
Behavioral: Blood Pressure Self-Monitoring — Participants engaged in blood pressure self-monitoring by measuring blood pressure twice daily and before and after exercise.
  Arms: EXERCISE+PEH

SUMMARY:
Sedentary (n=24) adults ≥18 yr with elevated BP to established hypertension were enrolled into this randomized clinical trial entitled, 'Blood Pressure UtiLizing Self-Monitoring after Exercise study or PULSE'. Participants were randomly assigned to either an exercise only (EXERCISE; n=12) or exercise plus BP self-monitoring (EXERCISE+PEH) (n=12) group. All participants participated in a 12 wk supervised moderate intensity aerobic exercise training program 40 min/d for 3 d/wk. In addition, they were encouraged to exercise at home ≥30 min/d for 1-2 d/wk. All participants self-monitored exercise with a traditional calendar recording method and heart rate (HR) monitor. In addition to traditional exercise self-monitoring (EXERCISE), individuals in the EXERCISE+PEH group were given a home BP monitor to assess home BP twice daily (in the morning upon awakening and in the evening) and prior to and after voluntary home exercise sessions. Resting BP, peak oxygen consumption (VO2peak), physical activity, dietary and salt intake, and antihypertensive medication adherence were measured before and after the 12 wk supervised exercise training program. In addition, integrated social-cognitive predictors of exercise that included questionnaires on exercise self-efficacy, barriers self-efficacy, outcome expectations for exercise, exercise intention, and affective responses to exercise were measured before and after the 12 wk supervised exercise training program. Four weeks following the completion of exercise training, self-reported exercise levels were assessed during a telephone interview in both groups. Among EXERCISE+PEH only, self-monitoring of BP was also self-reported during this telephone interview.

DETAILED DESCRIPTION:
A sub-study following the completion of the PULSE clinical trial investigated the reliability and time course of change of PEH during the 12-week exercise training program. Participants (n = 10) were PEH responders from the EXERCISE + PEH control arm who underwent 12 wk of supervised aerobic exercise training, 40 min/session at moderate-to-vigorous intensity for 3 d/wk. BP was assessed via a home BP monitor. PEH was calculated as post- minus pre-exercise BP for 36 sessions. To quantify the reliability of PEH, RMANCOVA and GRMANCOVA adjusted for pre-exercise BP derived the between-participant and measurement error variability that were used to calculate the intraclass correlation coefficient (ICC). The Akaike Information Criterion (AIC) compared the goodness-of-fit of the PEH models for each week of training.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 yr
* SBP ≥130 mmHg or DBP ≥80 mmHg or taking antihypertensive medication regardless of BP with a SBP <160 mmHg and DBP <100 mmHg
* Free of diagnosed cardiovascular, pulmonary, renal, metabolic, or other chronic diseases or depression
* Non-smokers for at least 6 mo prior to entry
* Consumed <2 alcoholic drinks daily
* Physically inactive defined as engaging in formal exercise ≤ 2d/wk.

Exclusion Criteria:

* Taking medications that influenced blood pressure such as inhaled or oral steroids, nonsteroidal anti-inflammatory agents, aspirin, and nutritional supplements with the exception of a 1-a-day vitamin, cold medications, and herbal supplements
* Osteoarthritis and orthopedic problems that compromised ability to exercise.
* Past medical history of cancer-related lymphedema
* Seeking to gain or lose weight
* Pregnant, lactating, or planning to become pregnant.
* Hormone-altering contraception administered in a bolus

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2016-10-28 (Actual); Primary Completion 2018-05-01 (Actual); Study Completion 2018-05-29 (Actual)

PRIMARY OUTCOMES:
Exercise Adherence | 12 weeks
  Exercise adherence to the 12 wk supervised portion of the aerobic exercise training program was calculated as the percent of supervised exercise sessions completed divided by the total number of supervised sessions possible (# of supervised sessions performed ÷ total number of possible supervised sessions X 100%). In this calculation, the total number of possible sessions was calculated as: 3 supervised exercise training days per wk for 12 wk = 36 sessions with a maximum possible adherence of 100% (e.g., 36÷36 X 100% =100%).
Blood Pressure Response to Exercise Training | 12 weeks
  The BP response to aerobic exercise training was calculated in two ways and in units 'mmHg': (1) in the laboratory (post training resting BP - pre training resting BP) during the control visits (Visits 1 or 2 vs. Visit 4 or 5); and (2) under ambulatory conditions (post training ambulatory BP - pre training ambulatory BP) following the control visits (Visits 1 or 2 vs. Visit 4 or 5) over the awake, sleep, and 19 hr.
Blood Pressure Response to Each Exercise Training Session | 12 weeks
  In the sub study analysis, the difference in post- minus pre-exercise resting BP from three weekly exercise sessions per participant for each week of training was calculated for both SBP and DBP (in units of 'mmHg')
Relative Change in Blood Pressure From Baseline for Each Exercise Session | 12 weeks
  The relative percent change in BP for each exercise session was calculated as post- minus pre-exercise BP divided by pre-exercise BP x 100%, for each exercise training session for both SBP and DBP. A negative percent change in SBP and/or DBP from baseline was deemed that postexercise hypotension occurred.
Reliability of Postexercise Hypotension | 12 weeks
  To quantify the reliability of postexercise hypotension, RMANCOVA and GRMANCOVA adjusted for pre-exercise BP derived the between-participant and measurement error variability that were used to calculate the intraclass correlation coefficient (unit-less)
Time Course of Change in the Magnitude of Postexercise Hypotension | 12 wk
  The Akaike Information Criterion (unit-less) was calculated to compare the goodness-of-fit of the postexercise hypotension models for each week of training and to determine the week of exercise training after which the the magnitude of reductions in SBP and DBP ceased to differ week-to-week.

SECONDARY OUTCOMES:
Exercise Training Characteristics: Frequency | 12 weeks
  Exercise training frequency (d/wk) was recorded for supervised, unsupervised, and supervised plus unsupervised exercise training over the course of 12wk.
Exercise Training Characteristics: Intensity | 12 weeks
  Exercise training intensity (%heart rate reserve) was recorded for supervised, unsupervised, and supervised plus unsupervised exercise training over the course of 12wk.
Exercise Training Characteristics: Time | 12 weeks
  Exercise training time (min) was recorded for supervised, unsupervised, and supervised plus unsupervised exercise training over the course of 12wk.
Exercise Training Characteristics: Type | 12 weeks
  Exercise training type (treadmill, cycle ergometer, elliptical) was recorded for unsupervised, and supervised plus unsupervised exercise training over the course of 12wk.
Integrated social-cognitive predictor of exercise | 12 weeks
  Participants were administered a validated questionnaire packet to assess whether EXERCISE and EXERCISE+PEH self-monitoring favorably modulated measures of integrated social-cognitive predictors of exercise (unitless).
Self Reported Physical activity | 12 weeks
  Participants were asked to maintain their usual lifestyle habits throughout study participation and were administered a validated questionnaire to assess self reported. physical activity (min).
Dietary Intake | 12 weeks
  Participants were asked to maintain their usual lifestyle habits throughout study participation and were administered a validated questionnaire to assess dietary intake (kcal/d).
Salt Intake | 12 weeks
  Participants were asked to maintain their usual lifestyle habits throughout study participation and were administered a validated questionnaire to assess salt intake (mg/d).
Antihypertensive Medication Adherence. | 12 weeks
  Participants taking antihypertensive medication were administered a validated questionnaire to assess antihypertensive medication adherence (%).

CONTACTS AND LOCATIONS:
Overall Officials: Linda S Pescatello, PhD, Principal Investigator — University of Connecticut

IPD SHARING:
Plan to Share IPD: Yes
All IPD data will be made available upon request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: All IPD data will be available upon request with no time limit.
Access Criteria: All IPD data will be shared and emailed to whoever requests it.